CLINICAL TRIAL: NCT00376337
Title: A Phase II, Multicenter, Randomized, Open-label, Active Controlled Study to Evaluate the Safety and Efficacy of Micafungin Salvage Mono-therapy Versus Active Control Intravenous Salvage Mono-therapy in Patients With Invasive Aspergillosis
Brief Title: Micafungin Salvage Mono-therapy in Invasive Aspergillosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to difficulties in recruitment and changes in standard care for invasive aspergillosis
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FG463-21-20
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2011-10

CONDITIONS: Invasive Aspergillosis
Keywords: Invasive Aspergillosis; Salvage Therapy; Micafungin
MeSH Terms: interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): infusion for 3-12 weeks
  Interventions: Drug: Systemic antifungal therapy
- 2 (Experimental): infusion for 3-12 weeks
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — IV
  Other Names: FK463
  Arms: 2
Drug: Systemic antifungal therapy — IV
  Arms: 1

SUMMARY:
To evaluate the efficacy and safety of micafungin in patients with proven invasive aspergillosis and who are refractory or intolerant to previous systemic antifungal therapy. To compare the efficacy and safety of the micafungin therapy with the active control arm

DETAILED DESCRIPTION:
This is a phase II, multicentre, prospective, active-controlled, open-label, 2:1 randomised and parallel group clinical study.

Patients will be stratified according to the baseline infection status and the baseline neutropenic status:

* Intolerant to previous antifungal therapy
* Refractory to previous antifungal therapy; progression of infection
* Refractory to previous antifungal therapy; failure to improve In case, criteria for both intolerant and refractory are fulfilled at the same time the patient will be considered as refractory.
* Neutropenic (absolute neutrophil count (ANC < 500 cells/mm3)
* Non neutropenic (ANC >= 500 cells/mm3)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with HSCT, acute leukaemia or myelodysplastic syndrome, with proven (probable only in case of pulmonary aspergillosis) invasive aspergillosis and refractory or intolerant to amphotericin B or voriconazole products

Exclusion Criteria:

* Patients with allergic bronchopulmonary aspergillosis, chronic pulmonary aspergillosis, aspergilloma, sinus aspergillosis or external otitis; patient with previous salvage therapy for the current episode of fungal infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Independent Data Review Board (IDRB) assessment of the overall success at the End of Treatment (EoT) defined as complete or partial clinical response. | Weeks 3-12

SECONDARY OUTCOMES:
Overall success at end of treatment | Weeks 3-12

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (43):
- Argentina (2):
  - Buenos Aires
  - La Plata
- Belgium (4):
  - Aalst
  - Brussels
  - Ghent
  - Leuven
- Brazil (10):
  - Belo Horizonte
  - Campinas
  - Curitiba
  - Goiânia
  - Ipatinga
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - Santo André
  - São Paulo
- Colombia (3):
  - Bogotá
  - Bucaramanga
  - Cali
- Croatia (2):
  - Rijeka
  - Zagreb
- Czechia (3):
  - Hradec Králové
  - Olomouc
  - Prague
- France (4):
  - Bobigny
  - Dijon
  - Paris
  - Pessac
- Germany (5):
  - Berlin
  - Bonn
  - Munich
  - Münster
  - Würzburg
- Budapest, Hungary
- Italy (3):
  - Monza
  - Pavia
  - Rozzano
- Poland (3):
  - Krakow
  - Lodz
  - Poznan
- Spain (3):
  - Madrid
  - Salamanca
  - Seville

REFERENCES:
- See also: Link to FDA website — http://www.accessdata.fda.gov/scripts/cder/drugsatfda